CLINICAL TRIAL: NCT05916131
Title: Pilot and Feasibility Trial of HypoPals, a Mobile Health Intervention for Improving Hypoglycemia Self-management in Type 1 Diabetes Adults Using Advanced Diabetes Technologies
Brief Title: Pilot Feasibility Study for HypoPals, a Mobile Health Program for Improving Hypoglycemia Management.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Yu Kuei Alex Lin, Associate Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00228484; 1K23DK129724-01 (NIH)
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes; Hypoglycemia
Keywords: hypoglycemia; mobile health technology; text messaging
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Adaptive randomization with minimization method will be conducted to ensure equal number of participants (n=10) will be randomized into the same number of the 4 experimental conditions (i.e., in 1:1:1:1 ratio). The randomization will be stratified based on whether the participant have severe hypoglycemia within the year or spending greater or equal to 1 percent of time in level 2 hypoglycemia on CGM, and the status of closed-loop pump use.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hypoglycemia Symptom Detection Training (Experimental): To provide Hypoglycemia Symptom Detection Training intervention.
  Interventions: Behavioral: Basic Education; Behavioral: Hypoglycemia Symptom Detection Training
- Education Plus (Experimental): To provide Education Plus intervention.
  Interventions: Behavioral: Basic Education; Behavioral: Education Plus
- Hypoglycemia Symptom Detection Training and Education Plus (Experimental): To provide both Hypoglycemia Symptom Detection Training and Education Plus interventions simultaneously.
  Interventions: Behavioral: Basic Education; Behavioral: Hypoglycemia Symptom Detection Training; Behavioral: Education Plus
- Usual Care (Other): Continuing usual care after basic education.
  Interventions: Behavioral: Basic Education

INTERVENTIONS:
Behavioral: Basic Education — 2-week text message intervention for providing knowledge about hypoglycemia management and prevention.
Behavioral: Hypoglycemia Symptom Detection Training — 10-week text message intervention for providing training on skills of detecting hypoglycemia symptoms.
  Arms: Hypoglycemia Symptom Detection Training; Hypoglycemia Symptom Detection Training and Education Plus
Behavioral: Education Plus — 10-week text message intervention for helping people consider how they think of hypoglycemia.
  Arms: Education Plus; Hypoglycemia Symptom Detection Training and Education Plus

SUMMARY:
A mobile health program "HypoPals", which incorporates data from continuous glucose monitoring systems (CGMs) and sends personalized text messages to help people sharpen their low blood sugar symptom detection skills, and help people consider how they think of low blood sugar, was devised. The goal of the current study is to make sure that HypoPals runs smoothly, users find the intervention useful, and the way the researchers conduct the final study will be correct (i.e., there is a need for 'pilot testing' the developed technology and research methods).

All participants will receive basic hypoglycemia education text messages, and then be randomized to one of the four experimental conditions: Hypoglycemia Symptom Detection Training, Education Plus, both Symptom Detection Training and Education Plus, and usual care. Participants may receive additional interventional text messages based on the experimental condition participants are assigned to.

The study may terminate after collecting sufficient data to evaluate the primary outcome (i.e., determining the number of participants recruited to reach 20 participants who complete the intervention).

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form
* Self-reported diagnosis of type 1 diabetes for at least 5 years
* Previous attendance of structured diabetes education program
* Using CGM greater or equal to (≥1) year
* Ongoing Dexcom CGM use time ≥70% based on CGM report at screening
* Have had experienced ≥1 episode of severe hypoglycemia in the past year while using CGMs or spending ≥1% of time in level 2 hypoglycemia at the time of pre-screening
* Using cellphone with functionality for sharing real-time data to Dexcom Clarity and receiving text messages
* Be able to communicate in English (spoken and written)
* Willing to comply with all study procedures including sharing CGM glucose information, receiving and reading intervention text messages, and completing study questionnaires

Exclusion Criteria:

* Active participation in clinical trials on diabetes/hypoglycemia interventions
* Pregnancy or planning for pregnancy within a year
* Untreated adrenal insufficiency or hypothyroidism
* Uncontrolled mental disorder or chronic cognitive dysfunctions (include but not limited to uncontrolled schizophrenia, depression and bipolar disorders; learning disability; active alcohol and substance dependence; dementia or cognitive impairment independent of hypoglycemia)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2025-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu Kuei Alex Lin, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hypoglycemia Symptom Detection Training | Education Plus | Hypoglycemia Symptom Detection Training and Education Plus | Usual Care
Started | 9 | 10 | 11 | 10
Completed 12 Week Intervention | 9 | 10 | 11 | 10
Completed ("Study Completion" meaning completed the intervention and all follow up appointments) | 9 | 10 | 10 | 10
Not Completed | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypoglycemia Symptom Detection Training | Education Plus | Hypoglycemia Symptom Detection Training and Education Plus | Usual Care | Total
Number analyzed (Participants) | 9 | 10 | 11 | 10 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: year] | 40 [31 to 49] | 43 [32 to 47] | 37 [28 to 43] | 42 [28 to 53] | 40 [30 to 46]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Men | 5 | 7 | 5 | 3 | 20
  Women | 4 | 3 | 6 | 6 | 19
  Prefer Not to Answer | 0 | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 1 | 5
  Not Hispanic or Latino | 8 | 8 | 10 | 9 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2 | 4
  White | 6 | 9 | 10 | 8 | 33
  More than one race | 2 | 1 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 10 | 11 | 10 | 40
Diabetes duration [Median (Inter-Quartile Range); unit: years] | 13 [8 to 23] | 16 [13 to 33] | 24 [16 to 29] | 24 [18 to 28] | 21 [13 to 26]
Hemoglobin A1C [Median (Inter-Quartile Range); unit: percent] | 6.2 [5.9 to 6.9] | 6.5 [6.0 to 6.9] | 6.4 [6.1 to 7.2] | 6.4 [5.6 to 7.1] | 6.4 [6.0 to 7.0]
Continuous Glucose Monitoring (CGM) use duration [Count of Participants; unit: Participants]
  1-2 years | 0 | 0 | 3 | 1 | 4
  3-6 years | 6 | 5 | 4 | 8 | 23
  More than 6 years | 3 | 5 | 4 | 1 | 13

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Recruited to Reach 20 Participants That Complete the Intervention
Description: This number will include participants that were enrolled and received part or all of the intervention.
Time Frame: Approximately 4.5 months
Population: Because this measure pertains to the study as a whole, regardless of arm, number of participants is not reported by arm.
Measure: Count of Participants; unit: Participants
Groups:
- Participants Recruited Who Completed the Intervention: All participants recruited who complete the intervention
Arm/Group | Participants Recruited Who Completed the Intervention
Number analyzed (Participants) | 20
Participants | 20

2. Secondary Outcome: Number of Potential Candidates Contacted During the Entire Recruitment Period
Description: This number includes all potential candidates for enrollment contacted during the entire recruitment period, regardless of whether or not they ultimately enrolled in the study.
Time Frame: Approximately 1 year (recruitment period)
Population: Total number of potential candidates who were contacted for potential enrollment, whether they were ultimately eligibility assessed/enrolled or not. Because this measure pertains to the study as a whole, regardless of arm, number of participants is not reported by arm.
Measure: Number; unit: Potential candidates
Groups:
- Patients Who Were Contacted: All patients who were contacted, whether eligibility assessed/enrolled or not.
Arm/Group | Patients Who Were Contacted
Number analyzed (Participants) | 227
Potential candidates | 227

3. Secondary Outcome: Percentage of Contacted Potential Candidates Being Eligible
Description: Percentage of contacted potential candidates who were eligibility-assessed and determined to be eligible for the study.
Time Frame: Approximately 1 year (recruitment period)
Population: All potential candidates who were contacted and completed the eligibility assessment for enrollment, regardless of whether or not they ultimately enrolled in the study.
Measure: Number; unit: Percent of assessed potential candidates
Groups:
- Potential Candidates Who Were Contacted and Screened for Potential Enrollment: All potential candidates who were contacted and completed the eligibility assessment
Arm/Group | Potential Candidates Who Were Contacted and Screened for Potential Enrollment
Number analyzed (Participants) | 114
Percent of assessed potential candidates | 35.1

4. Secondary Outcome: Rate of Participant Retention at 12 Weeks
Description: Number of participants who completed 12 weeks of the intervention
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Hypoglycemia Symptom Detection Training | Education Plus | Hypoglycemia Symptom Detection Training and Education Plus | Usual Care
Number analyzed (Participants) | 9 | 10 | 11 | 10
Participants | 9 | 10 | 11 | 10

5. Secondary Outcome: Rate of Participant Retention at 26 Weeks
Description: Number of participants who completed 26-week follow-up visit
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hypoglycemia Symptom Detection Training | Education Plus | Hypoglycemia Symptom Detection Training and Education Plus | Usual Care
Number analyzed (Participants) | 9 | 10 | 11 | 10
Participants | 9 | 10 | 10 | 10

6. Secondary Outcome: Rate of Participant Retention at 52 Weeks
Description: Number of participants who completed 52-week follow-up visit
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Hypoglycemia Symptom Detection Training | Education Plus | Hypoglycemia Symptom Detection Training and Education Plus | Usual Care
Number analyzed (Participants) | 9 | 10 | 11 | 10
Participants | 9 | 10 | 10 | 10

7. Secondary Outcome: Participants With Continuous Glucose Monitoring (CGM) Data Collected at 12 Weeks
Description: Percentage of participants whose CGM data was successfully collected at 12 weeks. Because percent is auto-calculated and displayed by ClinicalTrials.gov, the title has been simplified to reflect reporting number of participants for additional transparency.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Hypoglycemia Symptom Detection Training | Education Plus | Hypoglycemia Symptom Detection Training and Education Plus | Usual Care
Number analyzed (Participants) | 9 | 10 | 11 | 10
Participants | 9 | 10 | 11 | 10

8. Secondary Outcome: Participants With Continuous Glucose Monitoring (CGM) Data Collected at 26 Weeks
Description: Percentage of participants whose CGM data was successfully collected at 26 weeks. Because percent is auto-calculated and displayed by ClinicalTrials.gov, the title has been simplified to reflect reporting number of participants for additional transparency.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hypoglycemia Symptom Detection Training | Education Plus | Hypoglycemia Symptom Detection Training and Education Plus | Usual Care
Number analyzed (Participants) | 9 | 10 | 11 | 10
Participants | 9 | 10 | 11 | 10

9. Secondary Outcome: Participants With Continuous Glucose Monitoring (CGM) Data Collected at 52 Weeks
Description: Percentage of participants whose CGM data was successfully collected at 52 weeks. Because percent is auto-calculated and displayed by ClinicalTrials.gov, the title has been simplified to reflect reporting number of participants for additional transparency.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Hypoglycemia Symptom Detection Training | Education Plus | Hypoglycemia Symptom Detection Training and Education Plus | Usual Care
Number analyzed (Participants) | 9 | 10 | 11 | 10
Participants | 9 | 10 | 11 | 9

10. Secondary Outcome: Participants Reporting Reading Message Content at the End of the Intervention
Description: Assessed with a question adapted from mSustain questionnaire: "When you receive a HypoPals message, how much of it do you read?" Because percent is auto-calculated and displayed by ClinicalTrials.gov, the title has been simplified to reflect reporting number of participants for additional transparency.
Time Frame: 12 weeks
Population: The usual care group did not receive any intervention messages after completing the initial 2-week basic education.
Measure: Count of Participants; unit: Participants
Arm/Group | Hypoglycemia Symptom Detection Training | Education Plus | Hypoglycemia Symptom Detection Training and Education Plus
Number analyzed (Participants) | 9 | 10 | 11
Participants
  The whole message | 6 | 9 | 9
  About three-quarters of the message | 2 | 0 | 1
  About half of the message | 0 | 0 | 0
  About a quarter of the message | 0 | 1 | 1
  Not at all | 1 | 0 | 0

11. Secondary Outcome: Participants Finding Message Content Helpful (Positive) at the End of the Intervention
Description: Assessed with a study-purposed question: "Overall, HypoPals was helpful for me". Because percent is auto-calculated and displayed by ClinicalTrials.gov, the title has been simplified to reflect reporting number of participants for additional transparency.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Hypoglycemia Symptom Detection Training | Education Plus | Hypoglycemia Symptom Detection Training and Education Plus | Usual Care
Number analyzed (Participants) | 9 | 10 | 11 | 10
Participants
  Definitively | 4 | 3 | 1 | 3
  Between 'definitively' and 'somewhat' | 1 | 4 | 6 | 2
  Somewhat | 3 | 1 | 3 | 4
  Between 'somewhat' and 'not at all' | 1 | 1 | 0 | 0
  Not at all | 0 | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Hypoglycemia Symptom Detection Training | Education Plus | Hypoglycemia Symptom Detection Training and Education Plus | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 1/11 | 0/10
Other Adverse Events (participants affected / at risk) | 1/9 | 1/10 | 1/11 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypoglycemia Symptom Detection Training (N=9) | Education Plus (N=10) | Hypoglycemia Symptom Detection Training and Education Plus (N=11) | Usual Care (N=10)
Hospitalization due to Hypoglycemia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypoglycemia Symptom Detection Training (N=9) | Education Plus (N=10) | Hypoglycemia Symptom Detection Training and Education Plus (N=11) | Usual Care (N=10)
Hyperglycemia with/without confirmed ketosis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoglycemia requiring Emergency Medical Services (Endocrine disorders) | 0 (0) | 0 | 1 | 1 (1)
Food allergy (Immune system disorders) | 1 (1) | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 (0) | 0 | 0 | 1 (1)
Fibrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 | 0 | 1 (1)
Kidney stone (Renal and urinary disorders) | 0 (0) | 0 | 0 | 1 (1)
Papanicolaou smear abnormal (Reproductive system and breast disorders) | 0 (0) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
This is a pilot feasibility trial focused on the feasibility of running similar studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-06): https://cdn.clinicaltrials.gov/large-docs/31/NCT05916131/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT05916131/ICF_001.pdf